CLINICAL TRIAL: NCT03072329
Title: Neurostimulation in Pudendal Nerve Block: is That Really Necessary?
Brief Title: Neurostimulation in Pudendal Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital d'enfants Béchir-Hamza (Other)
Responsible Party: Principal Investigator, Dr Sonia ben khalifa (PhD), Head of Anesthesia and Intensive Care Department, Hôpital d'enfants Béchir-Hamza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNB-001
Record Dates: First submitted 2017-02-25; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Penile Surgery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pudendal nerve block (Experimental): Bilateral pudendal nerve block with the administration of 0.1 mL/kg Bupivacaïne 0.5%, regardless of neurostimulation response.
  Interventions: Procedure: Pudendal nerve block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Pudendal nerve block
Drug: Bupivacaine

SUMMARY:
The purpose of this study is to check whether the success rate of blind pudendal nerve block in penile surgery can be optimized by the search for a motor response during neurostimulation.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for elective penile surgery (hypospadias / circumcision)

Non-inclusion Criteria:

* Association to further peripheral nerve blocks required

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02-20 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Nerve block success | 15 minutes
  Nerve block success is defined by the absence of 20% increase in heart rate or systolic blood pressure baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Ben Khalifa Sonia, PhD, Principal Investigator
Locations (1):
- Hôpital d'Enfants Béchir Hamza, Bab Saadoun, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No